CLINICAL TRIAL: NCT01084850
Title: Corneal Endothelium Morphology and Central Thickness in Type II Diabetes Mellitus and Normal Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Jens christian Norregaard/Head of Department, Frederiksberg Hospital
Other Study IDs: FH5
Record Dates: First submitted 2010-02-25; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-01

CONDITIONS: Corneal Dystrophy
Keywords: Corneal endothelium; diabetes mellitus; corneal thickness
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes Type II: Patients with type 2 Diabetes Mellitus
- Control: Patients with no diabetes

SUMMARY:
The purpose of this study is to compare corneal endothelium morphology and central thickness in type II Diabetes Mellitus and normal subjects with special reference to glycemic status.

DETAILED DESCRIPTION:
Diabetes might influence the health of the corneal endothelium. Older studies have presented different results and the glycemic status of the patients have not been reported. In this study we examine the corneal endothelium morphology and central thickness in type II Diabetes Mellitus and normal subjects with modern specular microscopy. Each patient and control is examined once ("entry to study").

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes (diagnose confirmed by general practitioner)
* Controls with no diabetes (confirmed by blood testing).

Exclusion Criteria:

* Glaucoma
* Uveitis (current or previous)
* Corneal scaring
* Previous eye surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting Frederiksberg hospital for any reason
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Corneal endothelium cell number | 1 year
  The study is a cross-sectional study. We compare a cohort of patients with DM to a cohort with no DM. We examine each patient and control once. We call time of appointment or examination for "at entry to study".

SECONDARY OUTCOMES:
Corneal endothelium morphology | 1 year
  The size and hexagonality of the cells are analysed automaticly by computer recognizion.

CONTACTS AND LOCATIONS:
Overall Officials: Jens C Norregaard, MD, phd, Study Chair — Frederiksberg University Hospital, Eye Clinque
Locations (1):
- Frederiksberg University Eye Clinque, Frederiksberg, Frederiksberg, Denmark